CLINICAL TRIAL: NCT01278719
Title: 'The Factors Associated With the Formation of Nasal Polyp'
Brief Title: The Factors Associated With the Formation of Nasal polyp-a Case Control and Descriptive Study
Acronym: ACAAGSONP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karnataka Institute of Medical Sciences (Other)
Collaborators: Ministry of Science and Technology, India (Other Government); Applied Genetics (Industry); Lab Discoveries Ltd. (Industry)
Responsible Party: Principal Investigator, Manjunath dandinarasaiah, Department of ENT, Karnataka Institute of Medical Sciences
Other Study IDs: KIMSPGS412
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Nasal Polyp; Smoking; Rhinosinusitis; Allergic Rhinitis; Deviated Nasal Septum; ASA Intolerant Asthma
Keywords: Antrochoanal polyp; Ethmoidal polyp; Recurrence; Risk factors; Environmental factors; Gene expression; Micro array; Mutation
MeSH Terms: conditions — Nasal Polyps; Smoking; Rhinosinusitis; Rhinitis, Allergic; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Antrochaonal polyp; non recurrent type
- Antrochoanal polyp; recurrent type
- Ethmoidal polyp - non recurrent type
- Ethmoidal polyp - recurrent type

SUMMARY:
Nasal polyp is a significant health problem with a prevalence of 4%. It is increased in patients with asthma (7-15%), Cystic fibrosis (39-56%) or aspirin intolerance (36-96%).The quality of life (QOL) is worse than in patients suffering from hypertension, migraine, angina pectoris and head & neck cancer as per a previous study by Videler WJM et al.QOL is in comparison to chronic obstructive pulmonary disease.The reason why it develops in some and not in others remains unknown despite the disease being present for centuries.A definite relationship exists in patients with 'Sampter triad': Asthma, non steroidal anti-inflammatory drug sensitivity and nasal polyps. But not all patients with NSAID sensitivity have nasal polyps and vice verse.

Etiology is largely unknown despite the disease being present for centuries. Although the factors like wood stove exposure, smoking, allergic rhinitis, rhino sinusitis have been strongly implicated in literature from various studies, most data available is on ethmoidal polyps.The present study is an attempt to study the association of important risk factors with both antrochoanal(AC) and ethmoidal nasal polyps(EP).One study found that a significantly smaller proportion of the population with polyps were smokers compared to the unselected population (15% v/s 35%). But this is not confirmed by other studies.

Seven percent of asthma patients have nasal polyps and in non atopic asthma and late onset asthma, polyps are diagnosed more frequently (10-15%).Eosinophil numbers are significantly higher in nasal polyp tissue and further increased in patients with co-morbid asthma and aspirin sensitivity.

Nasal colonization in increased amounts was found by Staphylococcus aureus and presence of specific Immunoglobulin E directed against S.aureus enterotoxins was found. Rates of colonization and IgE presence in nasal polyp tissue were increased in subjects with nasal polyp associated with co-morbid asthma and aspirin sensitivity.

Nasal polyps are frequently found to run in families, suggesting a hereditary or with shared environmental factor. In the study by Rugina et al., more than half of 224 nasal polyp patients (52%) had a positive family history while the study by Greisener et.al, reported 14% of family history strongly suggesting hereditary factors in the pathogenesis of nasal polyps.

Some studies have found environmental factors like smoking and those using wood stove as a primary source of heating with the development of nasal polyps. The studies are contrasting.

There is presently a need of understanding the differences in the pathogenesis of antrochoanal polyp and ethmoidal nasal polyp clearly.There are hardly any concrete research performed on them to note the differences in the etiology and their pathogenesis. Hence the study is undertaken to extensively study the etiologies responsible for them and to note the differences.

DETAILED DESCRIPTION:
The present study involves two parts. A case control study wherein the association of nasal polyps with various risk factors like smoking, wood stove exposure, allergic rhinitis, non vegetarian diet intake, rhino sinusitis, deviated nasal septum, occupational dust exposure and eosinophilia.This will be studied individually for antrochoanal and ethmoidal nasal polyps.Again the same will be studied with respect to the recurrent and non recurrent polyps.

A descriptive study focuses on the nasal polyp occurrence with respect to the age, sex, religion, socioeconomic status, urban or rural preponderance,overcrowding, aspirin intolerance, family history etc.

The results will be studies after calculating the odds ratio and the chi square test for whatever data is available. Interpretation will be performed subsequently.

Gene expression profiling would be performed to study the differences in gene expression levels between AC and EP s with respect to risk factors and morphological characteristics.Mutational analysis will be performed to identify mutations in selected genes.

ELIGIBILITY:
Inclusion Criteria:

1. Antrochoanal and ethmoidal nasal polyps
2. Recurrent nasal polyps
3. Both infected and non infected polyps
4. Both eosinophilic and non eosinophilic polyps

Exclusion Criteria:

1. Exclusive neoplasms of nose and para nasal sinuses
2. Immunodeficiency status like HIV

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with nasal polyps attending Otorhinolaryngology outpatient department at the Karnataka institute of medical sciences, Hubli which is a tertiary care hospital situated in the north of Karnataka state in India.The hospital caters to all socioeconomic strata with vast diversities.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Association of the antrochoanal and ethmoidal polyps with smoking, wood stove exposure, allergic rhinitis, deviated nasal septum, rhino sinusitis, non vegetarian diet,eosinophilia and staphylococcus aureus in terms of the odds ratio. | 3 years
  Based on the questionnaire the patient will be evaluated for the presence of risk factors. Patient will be subjected to appropriate investigations like complete hemogram, absolute eosinophil count, contrast tomography scan of the paransal sinuses and serum IgE levels will be performed.An odds ratio will be calculated after taking appropriate controls in the ratio of 2:1.Significance levels will be calculated using Chi square test.
Gene expression profiling of Antrochoanal and Ethmoidal nasal polyps | 2yrs
  Three samples from each of the above three groups will be subjected to Microarray analysis. Differentially expressed genes will be selected and validation will be performed on 20 each of AC and EP groups.
Mutational analysis of Antrochoanal and Ethmoidal nasal polyps | 1year
  Once the genes have been identified based on Gene expression analysis, a few genes will be selected and studied for any possible mutations.

SECONDARY OUTCOMES:
Relationship of the nasal polyps with respect to the age, sex, religion, socioeconomic status, occupation, urban or rural preponderance, overcrowding and aspirin intolerance. | 3 years
  A descriptive analysis will be performed to know the relationship of the antrochoanal and ethmoidal polyps with the above factors in terms of the percentages and will be analyzed appropriately.
To study the cause for recurrence of Nasal polyps | 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Manjunath D Narasaiah, MS, Principal Investigator — Assistant Professor in ENT, Karnataka Institute of Medical Sciences, Hubli-580021, Karnataka, India
Locations (1):
- Department of Otorhinolaryngology, Karnataka Institute of Medical Sciences, Hubli, Karnataka, India

REFERENCES:
- [Background] Videler WJ, van Drunen CM, van der Meulen FW, Fokkens WJ. Radical surgery: effect on quality of life and pain in chronic rhinosinusitis. Otolaryngol Head Neck Surg. 2007 Feb;136(2):261-7. doi: 10.1016/j.otohns.2006.08.010. PMID 17275551
- [Result] Hedman J, Kaprio J, Poussa T, Nieminen MM. Prevalence of asthma, aspirin intolerance, nasal polyposis and chronic obstructive pulmonary disease in a population-based study. Int J Epidemiol. 1999 Aug;28(4):717-22. doi: 10.1093/ije/28.4.717. PMID 10480701
- [Result] Rugina M, Serrano E, Klossek JM, Crampette L, Stoll D, Bebear JP, Perrahia M, Rouvier P, Peynegre R. Epidemiological and clinical aspects of nasal polyposis in France; the ORLI group experience. Rhinology. 2002 Jun;40(2):75-9. PMID 12091997
- [Result] Kim J, Hanley JA. The role of woodstoves in the etiology of nasal polyposis. Arch Otolaryngol Head Neck Surg. 2002 Jun;128(6):682-6. doi: 10.1001/archotol.128.6.682. PMID 12049564
- [Result] Greisner WA 3rd, Settipane GA. Hereditary factor for nasal polyps. Allergy Asthma Proc. 1996 Sep-Oct;17(5):283-6. doi: 10.2500/108854196778662192. PMID 8922148
- [Result] Settipane GA, Chafee FH. Nasal polyps in asthma and rhinitis. A review of 6,037 patients. J Allergy Clin Immunol. 1977 Jan;59(1):17-21. doi: 10.1016/0091-6749(77)90171-3. PMID 833373